CLINICAL TRIAL: NCT03231176
Title: A Phase 2A, Single Arm, Multicentre, Study of Varlitinib Plus Capecitabine in Chinese Patients With Advanced or Metastatic Biliary Tract Cancer Who Progressed on at Least 1 Line of Systemic Therapy
Brief Title: Varlitinib Plus Capecitabine in Chinese Patients With Advanced or Metastatic Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASLAN001-008
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Biliary Tract Cancer
Keywords: Biliary Tract Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms
MeSH Terms: conditions — Biliary Tract Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Varlitinib and Capecitabine (Experimental)
  Interventions: Drug: Varlitinib; Drug: Capecitabine

INTERVENTIONS:
Drug: Varlitinib — oral tablets, twice daily
Drug: Capecitabine — oral tablets, twice daily for 2 weeks followed by a 1-week rest period in 3-week cycles

SUMMARY:
This protocol for Varlitinib is developed for the treatment of Biliary Tract Cancer. Varlitinib (also known as ASLAN001) is a small-molecule, adenosine triphosphate competitive inhibitor of the tyrosine kinases - epidermal growth factor receptor (EGFR), human epidermal growth factor receptor (HER)2, and HER4. Varlitinib may be beneficial to subjects with cancer by simultaneous inhibition of these receptors. The purpose of this study is to determine the safety and efficacy of Varlitinib in combination with capecitabine for the treatment of Biliary Tract Cancer. Eligible patients will receive Varlitinib plus capecitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed advanced (unresectable) or metastatic biliary tract cancer, including intrahepatic or extrahepatic cholangiocarcinoma, gallbladder cancer and carcinoma of the Ampulla of Vater. This includes clinical diagnosis of biliary tract cancer with histological confirmation of adenocarcinoma.
2. Patients who have received and failed one and only one prior line of systemic treatment or advanced or metastatic disease with radiologic evidence of disease progression. This prior line of systemic treatment must also contain gemcitabine
3. Patients with radiographically measurable disease based on RECIST v1.1.
4. Patients with no evidence of biliary duct obstruction, unless obstruction is controlled by local treatment or, in whom the biliary tree can be decompressed by endoscopic or percutaneous stenting with subsequent reduction in bilirubin to below 1.5 x upper level of normal (ULN).
5. Patients who are or older than 18 years of age and of or younger than 99 years of age at the time when written informed consent is obtained, and are able to understand and willing to sign the informed consent form.
6. Patients have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Patients with adequate organ and hematological function:

   1. Hematological function, as follows:

      * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
      * Platelet count ≥ 100 x 109/L
   2. Renal functions, as follows:

      * Estimated glomerular filtration rate or creatinine clearance > 50 mL/min/1.73m2
   3. Hepatic function, as follows:

      * Total bilirubin ≤ 1.5 x ULN
      * AST and ALT ≤ 5 x ULN

Exclusion Criteria:

1. Patients are currently on or have received anti-cancer therapy within the past 3 weeks.
2. Patients are currently on or have received radiation or local treatment within the past 3 weeks for the target lesion(s).
3. Patients have had major surgical procedures within 14 days prior to study entry.
4. Patients have a metastatic brain lesion(s), including asymptomatic and well controlled lesion(s).
5. Patients have malabsorption syndrome, diseases significantly affecting gastrointestinal function, resection of the stomach or small bowel, or difficulty in swallowing and retaining oral medications.
6. Patients have any history or presence of clinically significant condition which in the opinion of the Investigator could jeopardize the safety of the patient or the validity of the study results.
7. Patients have any history of other malignancy unless in remission for more than 1 year. (skin carcinoma and carcinoma-in-site of uterine cervix treated with curative intent is not exclusionary).
8. Female patients are pregnant or breast feeding.
9. Patients who been previously treated with varlitinib or have been previously treated with capecitabine as first line therapy for advanced or metastatic disease. For patients who have previously received capecitabine as radiosensitizer or as part of their adjuvant therapy and their disease has relapsed for more than 6 months after their last dose of capecitabine adjuvant therapy, their capecitabine therapy will not be considered as a line of systemic chemotherapy for metastatic/advanced disease, and thus they can participate in the study.
10. Patients have received any investigational drug (or have used an investigational device) within the last 14 days before receiving the first dose of study medication.
11. Patients have unresolved or unstable serious toxicity (≥CTCAE 4.03 Grade 2), with the exception of anemia, asthenia, and alopecia, from prior administration of another investigational drug and/or prior cancer treatment.
12. Patients have a known positive test for HIV, active hepatitis C, or hepatitis B infection with hepatitis B virus deoxyribonucleic acid exceeding 2000 IU/mL.
13. Patients have a known history of drug addiction within last 1 year, on the basis that there could be a higher risk of non-compliance to investigational product.
14. Patients need continuous treatment with proton pump inhibitors during the study period.
15. Patients have a baseline corrected QT interval QTc> 450 ms or patients with known long QT syndrome, torsade de pointes, symptomatic ventricular tachycardia, an unstable cardiac syndrome in the past 3 months before screening visit, > class 2 New York Heart Association heart failure, > grade 2 Canadian cardiovascular society angina pectoris, or receiving quinidine, procainamide, disopyramide, amiodarone, dronedarone, arsenic, dofetilide, or sotalol methadone.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Through study duration, estimated 2 years
  Objective Response Rate defined as the proportion of patients with a confirmed best response of partial response (PR) or complete response (CR), as defined by RECIST v1.1 criteria, based on an Independent Central Review (ICR) of radiological data.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Through study duration, estimated 2 years
  Progression Free Survival defined as the time from the start of treatment until the date of objective disease progression or death (by any cause in the absence of progression). Progression is defined in accordance with the RECIST v1.1 criteria and will be derived using data from the ICR.
Disease Control Rate (DCR) | Through study duration, estimated 2 years
  Disease control rate is defined as the number (%) of patients with a confirmed response of CR or PR, or with stable disease for a minimum of twelve weeks (- 5 days) from starting treatment.
Duration of Response (DoR) | Through study duration, estimated 2 years
  The Duration of Response is defined as the time from the date of first documented response until the date of documented disease progression or death in the absence of disease progression, in the subset of patient classified as confirmed responders for the assessment of ORR. The end of response should coincide with the date of disease progression or death from any cause used for the PFS endpoint. DoR will be calculated using the ICR data.
Overall Survival (OS) | Through study duration, estimated 2 years
  Overall Survival is defined as time from the start of treatment until death by any cause.
Safety and tolerability of varlitinib when combined with capecitabine | Through study duration, estimated 2 years
  Incidence of AEs, categorized in accordance to CTCAE 4.03, and changes from baseline in safety parameters

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - No.81 Hospital of The Chinese People's Liberation Army, Nanjing
  - There is 22 sites located in other cities of China, including Nanjing, Nanjing

IPD SHARING:
Plan to Share IPD: No